CLINICAL TRIAL: NCT03305380
Title: Radiomics to 1. Identify Patients at Risk for Developing Pneumonitis, 2. Differentiate Immune Checkpoint Inhibitor-induced Pneumonitis From Other Lung Inflammation and 3. Distinguish Tumour Pseudo-progression From Real Tumour Growth, in Patients With Non-small Cell Lung Cancer Treated With Anti-PD1 or Anti-PD-L1
Brief Title: Radiomics to Identify Patients at Risk for Developing Pneumonitis, Differentiate Immune Checkpoint Inhibitor-induced Pneumonitis From Other Lung Inflammation and Distinguish Tumour Pseudo-progression From Real Tumour Growth
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: BMS Radiomics
Record Dates: First submitted 2017-09-21; First posted 2017-10-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Stage IV Non-small Cell Lung Cancer
Keywords: anti-PD1; anti-PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a pulmonary event: (under anti-PD1 or anti-PD-L1) This is the first group of the retrospective part of the study.
  Interventions: Other: No interventions
- Patients without a pulmonary event: (under anti-PD1 or anti-PD-L1) This is the second group of the retrospective part of the study.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — As this is a patient registry, there are no interventions.

SUMMARY:
The investigators will develop a radiomics signature for immune checkpoint-induced pneumonitis in 40 patients with a pulmonary event under anti-PD1 or anti-PD-L1 (cases) and 40 patients without a pulmonary event under anti-PD1 or anti-PD-L1 (controls).

On the basis of the case-control study of patients treated with anti-PD1 or anti-PD-L1, they will further optimise the model using reinforcement machine learning. The model will then be validated in 300 prospective patients.

DETAILED DESCRIPTION:
Preliminary analyses on a dataset showed a clear distinction in radiomics features for patients with and without pneumonitis from anti-PD1 or anti-PD-L1. Prior experience of the investigators of training and validating radiomics signatures combined with their preliminary exploratory results presented here, will be used to develop a radiomics signature for immune checkpoint-induced pneumonitis in 40 patients with a pulmonary event under anti-PD1 or anti-PD-L1 (cases) and 40 patients without a pulmonary event under anti-PD1 or anti-PD-L1 (controls).

On the basis of the case-control study of patients treated with anti-PD1 or anti-PD-L1, the investigators will be able to further optimise the model using reinforcement machine learning. The model will then be validated in 300 prospective patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive standard anti-PD1 or anti-PD-L1 treatment in routine clinical practice for first or second line stage IV non-small cell lung cancer

Exclusion Criteria:

* The opposite of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive standard anti-PD1 or anti-PD-L1 treatment in routine clinical practice for first or second line stage IV non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Cause of pneumonitis | 6 months
  Determining cause of the pneumonitis by medical status of the patient

SECONDARY OUTCOMES:
Predictive accuracy of radiomics for determining the cause of pneumonitis | 6 months
  Three subgroups of immune checkpoint induced pneumonitis:
  1. Immune checkpoint-induced pneumonitis from tumour progression
  2. Immune checkpoint-induced pneumonitis from other types of pneumonitis
  3. Patients with interstitial lung disease that are at risk to develop immune checkpoint-induced pneumonitis and those who are not.
  Radiomics will be used to predict the cause of pneumonitis

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (2):
- Netherlands (2):
  - Zuyderland Medical Center, Heerlen
  - MUMC+, Maastricht

IPD SHARING:
Plan to Share IPD: No